CLINICAL TRIAL: NCT00307788
Title: The Association Amongst Acupuncture Analgesia, Expectancy, and Psychiatric Comorbidity in Patients With Low Back Pain
Brief Title: Acupuncture Analgesia in Relation to Psychiatric Comorbidity
Acronym: LBP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Ajay D. Wasan,M.D.,M.Sc., Psychiatrist, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2004P001139; P01AT002048-01 (NIH)
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Low Back Pain
Keywords: Psychiatric Comorbidity; Acupuncture; expectancy
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: acupuncture — acupuncture

SUMMARY:
It is our hypothesis that patient's expectations concerning treatment outcome will be influenced by their psychiatric symptoms, and that this expectancy will have a strong influence on the efficacy of acupuncture treatment to suppress experimentally induced pain. We will conduct a study, monitoring expectations but not manipulating them, in a cohort of patients with chronic low back pain.

DETAILED DESCRIPTION:
Specific Aim: To characterize subjective analgesia (behavioral effect) of different expectancy levels on verum and sham acupuncture treatment and the relative contribution of acupuncture treatment and expectancy to the resultant analgesia in healthy normals and in those with low back pain, controlling for psychiatric comorbidity.

Hypothesis 1: Patients with low back pain, low psychiatric comorbidity, and high expectations for acupuncture treatment will experience the same magnitude of acupuncture analgesia to thermal pain stimuli as healthy volunteers with high expectations for treatment.

Hypothesis 2: Patients with low back pain and high psychiatric comorbidity will experience less acupuncture analgesia compared to patients with low back pain and low psychiatric comorbidity, regardless of the level of expectations for acupuncture treatment.

Hypothesis 3: Patients with low back pain and high psychiatric comorbidity will have increased acupuncture placebo analgesia to thermal pain stimuli than both other groups.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers between 21 and 65 years of age with discogenic low back pain, either with or without radicular pain for more than three months, assessed by the treating physician with the use of imaging. Patients with discogenic low back are chosen in order to study a more uniform pain syndrome, a concern in pain medicine research [153]. Patients must have pain for at least three months because 90% of back pain resolves within three months of onset, and back pain beyond this time is more likely to remain chronic [156].
2. Average pain intensity of ≥4 on a scale from 0 to 10, because <4 is considered a level with acceptable pain and function
3. At least an 8th grade English-reading level; English can be a second language provided that the subjects feel they understand all the questions used in the assessment measures.
4. No long-acting opioids. Short acting opioids are acceptable, provided that subjects undergo a 7-10 day washout period. It is not possible to recruit an entirely opioid naïve population.
5. No prescription benzodiazepines.

Exclusion Criteria:

1. Any interventional procedure for low back or radicular pain two weeks prior to the study or during the two week study period, such as lumbar epidural steroids, nerve root blocks, or facet joint injections/ radiofrequency lesioning.
2. Having received acupuncture treatment before for any condition.
3. Back surgery in the previous 12 weeks, the intent to undergo back surgery during the study period, or any clinically unstable systemic illness that is judged to interfere with the trial.
4. Non-ambulatory status
5. History of cardiac or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome.
6. An inability to complete questionnaires accurately.
7. . Current opioid treatment through an intrathecal device
8. Cancer or other malignant disease, except carcinoma in situ of the skin or cervix

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pain relief | start and end
  %change in pain

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Wasan, M.D., MSc., Principal Investigator — Brigham and Women's Hospital; Bruce Rosen, MD, PhD, Study Director — Brigham and Womens Hospital
Locations (1):
- Pain Management Center, Chestnut Hill, Massachusetts, United States

REFERENCES:
- [Derived] Wasan AD, Kong J, Pham LD, Kaptchuk TJ, Edwards R, Gollub RL. The impact of placebo, psychopathology, and expectations on the response to acupuncture needling in patients with chronic low back pain. J Pain. 2010 Jun;11(6):555-63. doi: 10.1016/j.jpain.2009.09.013. Epub 2010 Jan 13. PMID 20075014